CLINICAL TRIAL: NCT07014423
Title: The Added Value of Three-dimensional Electroanatomic Mapping For Accurate Delivery Of Pulsed Field Ablation In The Pulmonary Veins Compared To Pulsed Field Ablation With Fluoroscopy And/Or Intracardiac Echocardiography Alone In The Treatment Of Atrial Fibrillation: MAP-PFA Study
Acronym: MAP-PFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL-009618
Record Dates: First submitted 2025-05-28; First posted 2025-06-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Electroanatomical mapping; Pulsed Field Ablation; Atrial Fibrillation; The FARAPULSE system; FARAWAVE catheter; FARAVIEW mapping software; Pulmonary vein isolation; Fluoroscopy; Intracardiac Echocardiography; High density mapping; Eccentricity Index
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is investigator-initiated, prospective, international, multicenter randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FARAVIEW group (Other): The FARAVIEW mapping software usage will be provided to this arm.
  Interventions: Procedure: The Pulsed Field Ablation to Isolate the Pulmonary Vein with the utilization of FARAVIEW mapping software.
- FARAWAVE Group (Other): This FARAVIEW mapping software will not be used in this arm.
  Interventions: Procedure: The Pulsed Field Ablation to Isolate the Pulmonary Vein without the utilization of FARAVIEW mapping software.

INTERVENTIONS:
Procedure: The Pulsed Field Ablation to Isolate the Pulmonary Vein with the utilization of FARAVIEW mapping software. — Pulmonary Vein Isolation with the additional use of the FARAVIEW mapping system (The additional mapping approach)
  Arms: FARAVIEW group
Procedure: The Pulsed Field Ablation to Isolate the Pulmonary Vein without the utilization of FARAVIEW mapping software. — Pulmonary Vein Isolation without the use of the FARAVIEW mapping system.
  Arms: FARAWAVE Group

SUMMARY:
This is a randomized control trial that aims to evaluate the added value of electro-anatomical mapping to improve the quality of pulse field ablation lesions during Atrial fibrillation ablation.

DETAILED DESCRIPTION:
This is a multi-center randomized control trial, aims to compare the symmetry and centricity of pulmonary veins antral ablation lesions during positioning the ablation catheter with versus without the use of the FARAVIEW mapping system. The trial will enroll patients with atrial fibrillation, who are planned to undergo atrial fibrillation pulsed field ablation ablation using FARAWAVE catheter (the standard ablation catheter without FARAVIEW mapping software utilization) and FARAVIEW catheter (the upgraded catheter with features to utilize the FARVIEW mapping software) during the period of 2025. A total of 32 patients will be randomized in 1:1 ratio to either group of the trial. The aim is to enroll 16 patients from each participating institution (i.e. UMCG and Erasmus UMC). All study candidates will be either assigned to FARAVIEW (Group 1) or FARAWAVE (Group 2). Both groups will undergo post ablation high density intracardiac mapping (e.g. voltage mapping) with the ORION mapping catheter, to assess the symmetry and centrality of the antral pulmonary veins' ablation lesions in relation to the pulmonary vein ostia. We propose an Eccentricity Index to compare and reflect the central location of the pulmonary veins' antral ablation lesions' margins relative to the pulmonary veins' ostia between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Atrial Fibrillation.
* Planned for ablation with Pulsed Field ablation technology.
* Able to consent for participation.

Exclusion Criteria:

-History of prior Atrial Fibrillation ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
The Eccentricity Index of the pulmonary veins' antral ablation lesions in both study groups. | Procedure Day

SECONDARY OUTCOMES:
The number of additional "touch-up" ablations needed according to the operator in both study groups after the initial ablation was concluded and post ablation map was performed. | Procedure Day

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Background] Roger A, Cottin Y, Bentounes SA, Bisson A, Bodin A, Herbert J, Maille B, Zeller M, Deharo JC, Lip GYH, Fauchier L. Incidence of clinical atrial fibrillation and related complications using a screening algorithm at a nationwide level. Europace. 2023 May 19;25(5):euad063. doi: 10.1093/europace/euad063. PMID 36938977
- [Background] Mark DB, Anstrom KJ, Sheng S, Piccini JP, Baloch KN, Monahan KH, Daniels MR, Bahnson TD, Poole JE, Rosenberg Y, Lee KL, Packer DL; CABANA Investigators. Effect of Catheter Ablation vs Medical Therapy on Quality of Life Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1275-1285. doi: 10.1001/jama.2019.0692. PMID 30874716
- [Background] Schaack D, Schmidt B, Tohoku S, Bordignon S, Urbanek L, Ebrahimi R, Hirokami J, Efe TH, Chen S, Chun KJ. Pulsed Field Ablation for Atrial Fibrillation. Arrhythm Electrophysiol Rev. 2023 Apr 14;12:e11. doi: 10.15420/aer.2022.45. eCollection 2023. PMID 37427302
- [Background] Kuwahara T. Intracardiac Echocardiography in Catheter Ablation for Atrial Fibrillation: It Is Better to See What You Are Doing? J Atr Fibrillation. 2015 Apr 30;7(6):1215. doi: 10.4022/jafib.1215. eCollection 2015 Apr-May. PMID 27957164
- [Background] Rolf S, Hindricks G, Sommer P, Richter S, Arya A, Bollmann A, Kosiuk J, Koutalas E. Electroanatomical mapping of atrial fibrillation: Review of the current techniques and advances. J Atr Fibrillation. 2014 Dec 31;7(4):1140. doi: 10.4022/jafib.1140. eCollection 2014 Dec. PMID 27957132
- [Background] Nedios S, Sommer P, Bollmann A, Hindricks G. Advanced Mapping Systems To Guide Atrial Fibrillation Ablation: Electrical Information That Matters. J Atr Fibrillation. 2016 Apr 30;8(6):1337. doi: 10.4022/jafib.1337. eCollection 2016 Apr-May. PMID 27909489
- [Background] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321
- [Background] Reddy VY, Koruth J, Jais P, Petru J, Timko F, Skalsky I, Hebeler R, Labrousse L, Barandon L, Kralovec S, Funosako M, Mannuva BB, Sediva L, Neuzil P. Ablation of Atrial Fibrillation With Pulsed Electric Fields: An Ultra-Rapid, Tissue-Selective Modality for Cardiac Ablation. JACC Clin Electrophysiol. 2018 Aug;4(8):987-995. doi: 10.1016/j.jacep.2018.04.005. Epub 2018 May 11. PMID 30139499
- [Background] Badertscher P, Knecht S, Rosso R, Krisai P, Spreen D, Katic J, Du Fay de Lavallaz J, Sticherling C, Kuhne M. How to perform pulmonary vein isolation using a pentaspline pulsed field ablation system for treatment of atrial fibrillation. Heart Rhythm. 2025 Jan;22(1):69-79. doi: 10.1016/j.hrthm.2024.06.058. Epub 2024 Jul 2. No abstract available. PMID 38964447
- [Background] Goto K, Miyazaki S, Negishi M, Ikenouchi T, Yamamoto T, Kawamura I, Nishimura T, Takamiya T, Tao S, Takigawa M, Sasano T. Distribution of antral lesions with the novel size-adjustable cryoballoon for pulmonary vein isolation and the differences based on left atrial remodeling. J Cardiovasc Electrophysiol. 2024 Nov;35(11):2099-2108. doi: 10.1111/jce.16415. Epub 2024 Aug 21. PMID 39169533
- [Background] Rems L, Rainot A, Wiczew D, Szulc N, Tarek M. Cellular excitability and ns-pulsed electric fields: Potential involvement of lipid oxidation in the action potential activation. Bioelectrochemistry. 2024 Feb;155:108588. doi: 10.1016/j.bioelechem.2023.108588. Epub 2023 Oct 12. PMID 37879163
- [Background] Kotnik T, Rems L, Tarek M, Miklavcic D. Membrane Electroporation and Electropermeabilization: Mechanisms and Models. Annu Rev Biophys. 2019 May 6;48:63-91. doi: 10.1146/annurev-biophys-052118-115451. Epub 2019 Feb 20. PMID 30786231
- [Background] Lee RC. Cell injury by electric forces. Ann N Y Acad Sci. 2005 Dec;1066:85-91. doi: 10.1196/annals.1363.007. PMID 16533920
- [Background] Asad ZUA, Yousif A, Khan MS, Al-Khatib SM, Stavrakis S. Catheter Ablation Versus Medical Therapy for Atrial Fibrillation: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Circ Arrhythm Electrophysiol. 2019 Sep;12(9):e007414. doi: 10.1161/CIRCEP.119.007414. Epub 2019 Aug 21. PMID 31431051
- [Background] Elsheikh S, Hill A, Irving G, Lip GYH, Abdul-Rahim AH. Atrial fibrillation and stroke: State-of-the-art and future directions. Curr Probl Cardiol. 2024 Jan;49(1 Pt C):102181. doi: 10.1016/j.cpcardiol.2023.102181. Epub 2023 Oct 31. PMID 37913929
- [Background] Wu J, Nadarajah R. The growing burden of atrial fibrillation and its consequences. BMJ. 2024 Apr 17;385:q826. doi: 10.1136/bmj.q826. No abstract available. PMID 38631724
- [Background] Wyndham CR. Atrial fibrillation: the most common arrhythmia. Tex Heart Inst J. 2000;27(3):257-67. PMID 11093410
- [Background] Ko D, Chung MK, Evans PT, Benjamin EJ, Helm RH. Atrial Fibrillation: A Review. JAMA. 2025 Jan 28;333(4):329-342. doi: 10.1001/jama.2024.22451. PMID 39680399